CLINICAL TRIAL: NCT07052903
Title: TRITON-CM: A Phase 3 Global, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Nucresiran in Patients With Transthyretin-Mediated Amyloidosis With Cardiomyopathy (ATTR Amyloidosis With Cardiomyopathy)
Brief Title: TRITON-CM: A Study to Evaluate Nucresiran in Patients With Transthyretin Amyloidosis With Cardiomyopathy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-TTRSC04-003; 2024-519917-72-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Amyloidosis With Cardiomyopathy
Keywords: ATTR-CM; ATTR amyloidosis with cardiomyopathy; ATTR; Heriditary ATTR; hATTR; Wild-type ATTR; wATTR; Cardiomyopathy; Amyloidosis; TTR; Transthyretin; TTR-mediated amyloidosis; RNAi; RNAi therapeutic; TTR cardiomyopathy; V122i; TTR amyloidosis
MeSH Terms: conditions — Cardiomyopathies; Amyloidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive placebo administered subcutaneously (SC) once every 6 months (q6M) during the double-blind (DB) period, followed by nucresiran 300 mg administered SC q6M during the open-label extension (OLE) period.
  Interventions: Drug: Nucresiran; Drug: Sterile Normal Saline (0.9% NaCl)
- Nucresiran 300 mg (Experimental): Participants will receive nucresiran 300 mg administered SC Q6M during the DB period, followed by nucresiran 300 mg administered SC q6M during the OLE period.
  Interventions: Drug: Nucresiran

INTERVENTIONS:
Drug: Nucresiran — Nucresiran 300 mg administered SC q6M
  Other Names: ALN-TTRSC04
Drug: Sterile Normal Saline (0.9% NaCl) — Sterile Normal Saline (0.9% NaCl) administered SC once q6M
  Arms: Placebo

SUMMARY:
The purpose of this study is to:

* Evaluate the efficacy of nucresiran compared to placebo on reducing all-cause mortality and cardiovascular (CV) events
* Evaluate the efficacy of nucresiran compared to placebo on additional assessments of CV events and/or death
* Evaluate the efficacy of nucresiran compared to placebo on patient-reported health status and health-related quality of life

ELIGIBILITY:
Inclusion Criteria

* Has documented diagnosis of ATTR amyloidosis with cardiomyopathy including those with hereditary ATTR (hATTR) or wild-type ATTR (wATTR) amyloidosis.
* Has medical history of heart failure (HF) with at least 1 prior hospitalization for HF or signs and symptoms that require treatment with a diuretic.
* Has screening N-terminal prohormone B-type natriuretic peptide (NT-proBNP) >300 ng/L and <8500 ng/L; In patients with permanent or persistent atrial fibrillation, screening NT-proBNP >600 ng/L and <8500 ng/L.
* Patients may be receiving approved TTR stabilizers for ATTR amyloidosis (eg, tafamidis, acoramidis) and may be receiving background therapy for HF at the discretion of the Investigator.

Exclusion Criteria

* Has New York Heart Association (NYHA) Class IV HF; or NYHA Class III heart failure AND ATTR Amyloidosis Disease Stage 3.
* Has a polyneuropathy disability (PND) Score IIIa, IIIb, or IV.
* Has an estimated glomerular filtration rate eGFR of <30 mL/min/1.73m^2 at screening.
* Has received prior or currently receiving TTR-lowering therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2030-05-28 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of all-cause mortality and recurrent cardiovascular [CV] events (CV hospitalizations and urgent heart failure [HF] visits) | Baseline to end of double-blind period (estimated 32 months, maximum 5 years)
  All-cause mortality and recurrent CV events (CV hospitalizations and urgent HF visits) will be compared between treatment groups using an Andersen-Gill model.

SECONDARY OUTCOMES:
Time to first CV event (CV hospitalizations and urgent HF visits) or all-cause mortality | Baseline to end of double-blind period (estimated 32 months, maximum 5 years)
All-cause mortality | Baseline to end of double-blind period (estimated 32 months, maximum 5 years)
Recurrent CV events (CV hospitalizations and urgent HF visits) | Baseline to end of double-blind period (estimated 32 months, maximum 5 years)
Change from baseline in Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ-OS) | Baseline to Month 30
  The KCCQ is a 23-item self-administered questionnaire quantifying 6 domains (symptoms, physical function, quality of life, social limitation, self-efficacy, and symptom stability) and 2 summary scores (clinical and overall summary [OS]). Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (57):
- United States (13):
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Brandon, Florida
  - Clinical Trial Site, Gainesville, Georgia
  - Clinical Trial Site, Tucker, Georgia
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Manhasset, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
- Clinical Trial Site, Rosario, S, Argentina
- Australia (2):
  - Clinical Trial Site, Box Hill, Victoria
  - Clinical Trial Site, Joondalup, Western Australia
- Clinical Trial Site, Braunau am Inn, Austria
- Clinical Trial Site, Roeselare, Belgium
- Clinical Trial Site, Rio de Janeiro, Brazil
- China (5):
  - Clinical Trial Site, Fuzhou
  - Clinical Trial Site, Guangzhou
  - Clinical Trial Site, Hangzhou
  - Clinical Trial Site, Shanghai
  - Clinical Trial Site, Shenzhen
- France (3):
  - Clinical Trial Site, Rouen
  - Clinical Trial Site, Strasbourg
  - Clinical Trial Site, Toulouse
- Germany (2):
  - Clinical Trial Site, Leipzig, Saxony
  - Clinical Trial Site, Dresden
- Israel (2):
  - Clinical Trial Site, Be’er Ya‘aqov
  - Clinical Trial Site, Petah Tikva
- Clinical Trial Site, Ancona, Italy
- Japan (5):
  - Clinical Trial Site, Fukuoka
  - Clinical Trial Site, Kobe
  - Clinical Trial Site, Nankoku
  - Clinical Trial Site, Okayama
  - Clinical Trial Site, Sapporo
- New Zealand (2):
  - Clinical Trial Site, Christchurch, CAN
  - Clinical Trial Site, Hamilton, WKO
- Clinical Trial Site, Ålesund, Norway
- Spain (9):
  - Clinical Trial Site, Jaén, Andalusia
  - Clinical Trial Site, Bilbao, Basque Country
  - Clinical Trial Site, Barcelona, B
  - Clinical Trial Site, Vigo, Galicia
  - Clinical Trial Site, Huelva, H
  - Clinical Trial Site, Palma de Mallorca, IB
  - Clinical Trial Site, Madrid, Madrid
  - Clinical Trial Site, Valencia, V
  - Clinical Trial Site, Pamplona
- Switzerland (4):
  - Clinical Trial Site, Basel, Canton of Basel-City
  - Clinical Trial Site, Bern
  - Clinical Trial Site, Geneva
  - Clinical Trial Site, Lucerne
- Clinical Trial Site, Taichung, Taiwan
- United Kingdom (3):
  - Clinical Trial Site, Birmingham, BIR
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.